CLINICAL TRIAL: NCT02955810
Title: Phase Ib Study of Weekly Cyclophosphamide-Bortezomib-Dexamethasone (CyBorD) With Daratumumab (DARA) in Transplant Eligible Patients With Newly Diagnosed Multiple Myeloma (MM): "The CyBorD-DARA Study"
Brief Title: Cyclophosphamide-Bortezomib-Dexamethasone (CyBorD) With Daratumumab (DARA)
Acronym: CyBorD-Dara
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Cancer Trials Ireland (Network)
Responsible Party: Principal Investigator, Michael O'Dwyer, Professor of Medicine, National University of Ireland, Galway, Ireland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-BCNI-001
Record Dates: First submitted 2016-10-18; First posted 2016-11-04 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed; Treatment Naiive
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Cyclophosphamide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CyBorD-DARA (Experimental)
  Interventions: Drug: Daratumumab; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab
  Other Names: Darzalex
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Bortezomib
  Other Names: Velcade
Drug: Dexamethasone

SUMMARY:
This study is a Phase Ib open label, single arm, adaptive multicentre trial. Patients with newly diagnosed Multiple Myeloma (MM) will be treated with Cyclophosphamide-Bortezomib-Dexamethasone (CyBorD) in combination with Daratumumab (DARA).

The safety profile of daratumumab to date, which does not appear to overlap with those known for approved agents, combined with its distinct MoA, suggest that the therapeutic profile of daratumumab combined with various backbone regimens may improve the treatment effect of these regimens. Additionally, daratumumab as a single agent may prolong the progression free interval for these patients. Based on the potential for cyclophosphamide to enhance ADCP, there is a strong rationale to combine DARA with a cyclophosphamide, bortezomib containing regimen. This will be the first clinical trial to explore the feasibility of combining daratumumab with a cyclophosphamide containing backbone induction regimen and if successful will provide the rationale for larger studies exploring the efficacy of this combination in greater detail.

DETAILED DESCRIPTION:
The study will consist of 2 phases:

* The Screening Phase will extend up to 28 days prior to Cycle 1, Day 1.
* The Treatment Phase will be conducted in 2 parts and will extend from Cycle 1 Day 1 until treatment discontinuation.

Treatment Phase, Part 1: Induction/Transplantation/Consolidation Phase. The consolidation phase of treatment will begin approximately 30-60 days after Autologous Stem Cell Transplantation (ASCT), when the patient has recovered sufficiently and engraftment is complete.

Treatment Phase, Part 2: Maintenance Phase treatment until a maximum duration of 2 years, documented disease progression, death, loss to follow-up, or withdrawal of consent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study.
* Patient must be between 18 and <70 years of age.
* Patient must have documented diagnosis of multiple myeloma requiring treatment as per IMWG updated criteria for the diagnosis of multiple myeloma and measurable disease as defined by:

  * Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma
  * Measurable disease as defined by any of the following:
  * IgG multiple myeloma: serum monoclonal paraprotein (M-protein) level

    ≥1.0g/dl or urine M-protein level ≥200mg/24 hours; or
  * IgA, IgE, IgD or IgM multiple myeloma: serum M-protein level ≥0.5g/dl or urine M-protein level ≥200mg/24 hours; or
  * Light chain multiple myeloma without measurable disease in the serum or the urine: serum immunoglobulin free light chain ≥10mg/dl and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Newly diagnosed patient eligible for high dose therapy and autologous stem cell transplantation.
* Patient must have an ECOG performance status score of 0-2.
* Patient must have pre-treatment clinical laboratory values meeting the following criteria during the Screening Phase:

  * Haemoglobin ≥7.5g/dl (≥5mmol/l); prior red blood cell [RBC] transfusion or recombinant human erythropoietin use is permitted);
  * absolute neutrophil count (ANC) ≥1.0x109/l (GCSF is permitted);
  * AST ≤ 2.5 x upper limit of normal (ULN);
  * ALT ≤ 2.5 x ULN;
  * total bilirubin ≤ 1.5 x ULN (except in patients with congenital bilirubinaemia, such as Gilbert syndrome, direct bilirubin ≤ 1.5 x ULN);
  * calculated creatinine clearance ≥40ml/min/1.73m2;
  * corrected serum calcium ≤ 14mg/dl (<3.5mmol/l); or free ionized calcium ≤6.5mg/dl (≤1.6mmol/l);
  * platelet count ≥70x109/l for patients in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count >50x109/l (transfusions are not permitted to achieve this minimum platelet count).
* Patients who are women of child-bearing potential or male partners of women of childbearing potential must agree to use adequate contraception methods from signing of the informed consent form until at least 4 months after the last study drug administration.
* Childbearing potential is defined as any woman who has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally post-menopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months). The investigator or a designated associate is required to advise the patient how to achieve adequate birth control. Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include: combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal) progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable), intrauterine device (IUD), intrauterine hormone -releasing system (IUS), bilateral tubal occlusion, successfully vasectomised partner and sexual abstinence. In addition, the use of condoms by patients or their partners is required unless the woman has had a hysterectomy. Contraception will start 4 weeks before the start of therapy, will continue during therapy including dose interruptions and for 4 months after the last dose of any component of the treatment regimen.
* A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 10 to 14 days prior to first dose and the second within 24 hours prior to first dose.
* Patient must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Patient has received daratumumab or other anti-CD38 therapies previously.
* Patient has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma. Monoclonal gammopathy of undetermined significance is defined by presence of serum M-protein < 3g/dl; absence of criteria consistent with active/symptomatic multiple myeloma as per IMWG criteria. Smoldering multiple myeloma is defined as asymptomatic multiple myeloma with absence of related organ or tissue impairment (ROTI) end organ damage.
* Patient has a diagnosis of Waldenstrom's macroglobulinemia or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
* Patient has prior or current systemic therapy or stem cell transplantation for any plasma cell dyscrasia, with the exception of an emergency use of a short course (equivalent of dexamethasone 40mg/day for a maximum 4 days) of corticosteroids before treatment.
* Patient has peripheral neuropathy or neuropathy grade 2 or higher, as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
* Patient has had any prior or concurrent invasive malignancy (other than multiple myeloma) within 5 years of screening period except adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, localized prostate adenocarcinoma diagnosed ≥3 years and without evidence of biochemical failure, or other cancer for which the patient has undergone potentially curative therapy and has no evidence of that disease for ≥10 years.
* Patient has had radiation therapy within 14 days prior to start of study treatment.
* Patient has had plasmapheresis within 28 days of registration.
* Patient is exhibiting clinical signs of meningeal involvement of multiple myeloma.
* 10. a) Patient has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and patients must be excluded if FEV1 < 50% of predicted normal.

  b) Patient has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. (Note that patients who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
* Patient is known to be seropositive for or active human immunodeficiency virus (HIV) or known to have active hepatitis B or hepatitis C.
* Patient has any concurrent medical or psychiatric condition or disease (e.g. active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
* Patient has clinically significant cardiac disease, including:

  * myocardial infarction within 1 year before registration, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (e. g. unstable angina, congestive heart failure, New York Heart Association Class IIIIV), OR
  * cardiac arrhythmia (NCI-CTCAE Version 4.0 Grade ≥ 2) or clinically significant ECG abnormalities, and
  * screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
* Patient has known allergies, hypersensitivity, or intolerance to boron or mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the DARA Investigator's Brochure), or known sensitivity to mammalian-derived products.
* Patient has plasma cell leukaemia (according to WHO criterion: ≥20% of cells in the peripheral blood with an absolute plasma cell count of more than 2x109/l) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Patient is known or suspected of not being able to comply with the study protocol (e.g. because of alcoholism, drug dependency, or psychological disorder). Patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g. compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Patient is a woman who is pregnant, or breast-feeding, or planning to become pregnant while participating in this study or within 4 months after the last dose of any component of the treatment regimen. Or, patient is a man who plans to father a child while included in this study or within 4 months after the last dose of any component of the treatment regimen.
* Patient has had major surgery within 2 weeks before registration or will not have fully recovered from surgery, or has surgery planned during the time the patient is expected to participate in the study. Kyphoplasty is not considered major surgery.
* Patient has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before registration or is currently enrolled in an interventional investigational study.
* Patient has contraindication to the use of any components of the treatment regimen, per the Summary of Product Characteristics.
* Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
MTD | 15 months
  To determine the Maximum Tolerated Dose (MTD) for cyclophosphamide and bortezomib that can be safely administered with DARA.
The rate of Complete Response (CR) post Autologous Stem Cell Transplantation (ASCT) | 42 months
  Efficacy assessed by the rate of Complete Response (CR) post Autologous Stem Cell Transplantation (ASCT)

SECONDARY OUTCOMES:
Safety and Tolerability as assessed by adverse events | 42 months
  Safety and Tolerability will be assessed by standard clinical and laboratory tests. Adverse event grades will be determined by the NCI CTCAE v4.03
Complete Response Rate at the end of induction, ASCT, consolidation and maintenance | 42 months
Best Overall Response | 42 months
Minimal Residual Disease (MRD) negative rate at the end of induction, ASCT, consolidation and maintenance | 42 months
Progression Free Survival (PFS) at the end of maintenance phase | 42 months
Overall Survival (OS) at the end of maintenance phase | 42 months
Clinical Benefit Rate (CBR) | 42 months

CONTACTS AND LOCATIONS:
Locations (1):
- Galway University Hospital, Galway, Ireland

REFERENCES:
- [Derived] O'Dwyer M, Henderson R, Naicker SD, Cahill MR, Murphy P, Mykytiv V, Quinn J, McEllistrim C, Krawczyk J, Walsh J, Lenihan E, Kenny T, Hernando A, Hirakata G, Parker I, Kinsella E, Gannon G, Natoni A, Lynch K, Ryan AE. CyBorD-DARA is potent initial induction for MM and enhances ADCP: initial results of the 16-BCNI-001/CTRIAL-IE 16-02 study. Blood Adv. 2019 Jun 25;3(12):1815-1825. doi: 10.1182/bloodadvances.2019000010. PMID 31201169